CLINICAL TRIAL: NCT03931863
Title: The Effect of Ondansetron on Spinal Anesthesia in Caesarean Section
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aretaieion University Hospital (Other)
Collaborators: University of Athens (Other)
Responsible Party: Principal Investigator, Stavroula Karachanidi, Principal Investigator, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 124/17-04-2019
Record Dates: First submitted 2019-04-24; First posted 2019-04-30 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Hypotension
Keywords: ondansetron
MeSH Terms: conditions — Hypotension | interventions — Ondansetron; onda cryl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All solutions will be prepared by an independent researcher who will not be further involved in the study eg data collecting or analyzing them. All solutions will look identical to the anesthetist who will administer them to the patients.Apart from the anesthetist, the surgery staff and the researchers recording the measurements will not know the therapeutic intervention team in which each patient has been randomized.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Active Comparator): Intravenous administration of ondansetron 4mg diluted in 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Interventions: Drug: Ondansetron 4mg
- Group B (Active Comparator): Intravenous administration of ondansetron 8mg diluted in 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Interventions: Drug: Ondansetron 8mg
- Group C (Placebo Comparator): Intravenous administration of 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Interventions: Drug: 100ml normal saline 0.9 percent

INTERVENTIONS:
Drug: Ondansetron 4mg — Intravenous administration of ondansetron 4mg diluted in 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Other Names: Onda
  Arms: Group A
Drug: Ondansetron 8mg — Intravenous administration of ondansetron 8mg diluted in 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Other Names: Onda
  Arms: Group B
Drug: 100ml normal saline 0.9 percent — Intravenous administration of 100ml of normal saline 0.9 percent within 10 minutes prior to spinal anesthesia.
  Other Names: N/S 0.9 percent
  Arms: Group C

SUMMARY:
The purpose of this study is to compare the administration of two different doses of ondansetron to placebo to prevent hypotension and bradycardia following spinal anaesthesia. Apart from haemodynamic parameters (blood pressure and heart rate),characters of the spinal blockage (time of onset and regression) will be recorded too.

DETAILED DESCRIPTION:
The day before surgery the procedure will be explained to the patient and the written consent will be obtained. In the operating room, intraoperative monitoring will include electrocardiography (ECG), noninvasive blood pressure, oxygen saturation by pulse oximetry (SpO2) and heart rate (HR). Two peripheral intravenous catheters wil be placed for fluid replacement and administration of drugs.

Participants will be randomly assigned to one of the following groups:

Group A: Women will receive 4 milligrams (mg) of ondansetron diluted in 100 milliliters (ml) of normal saline 0.9 percent 10 minutes before spinal anaesthesia

Group B:Women will receive 8 mg of ondansetron diluted in 100ml of normal saline 0.9 percent 10 minutes before spinal anaesthesia

Group C:Women will receive 100ml of normal saline 0.9 percent 10 minutes before spinal anaesthesia

Subsequently, after receiving 500ml of colloid solution, spinal anesthesia will be performed at level L3-L4 or L4-L5 in the vertebral space with 1.6ml of 0.75 percent ropivacaine and 15mcg of fentanyl, using a 27-gauge pencil point spinal needle with patients in a left lateral position. After subarachnoid infusion, participants will be placed supine with left uterine displacement and anesthetic and motor blockage will be evaluated every one minute until anesthetic blockage reaches the level of T4 neurotome and the motor block becomes complete (Bromage grade 3). This time will be called Time to max effect (Tmax).

Hypotension, defined as systolic blood pressure below 100 millimeters of Mercury (mmHg), will be treated using 5mg ephedrine if the heart rate is less than 100 beats per minute or with 20mcg of phenylephrine if the heart rate is greater than 100 beats per minute. Bradycardia, defined as a fall in heart rate below 60 beats per minute will be treated with atropine (0.6mg).

Immediately after the delivery of the neonate, all women will receive a solution of oxytocin (20 units) intravenously. Half an hour before the end of the procedure they will receive an additional 1g of paracetamol and 75mg of diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* Physical status according to American Society of Anesthesiologists (ASA) I-II
* Singleton pregnant women in full term pregnancy
* Patients scheduled for cesarean section
* Height 158cm-170cm

Exclusion Criteria:

* patient's own refusal
* contraindications to spinal anesthesia (coagulation disorders, inflammation at the puncture site, allergy to local anesthetics)
* ondansetron allergy
* body mass index> 33kg / m^2
* height <158cm, or> 170cm
* hypertensive disorders of pregnancy
* cardiovascular disease
* receiving selective serotonin reuptake inhibitors (SSRI's) or treatment for migraine
* placenta previa.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure during cesarean section | 60 minutes
  every one minute after spinal anaesthesia and every five minutes after the delivery of the neonate until the end of the surgery
Change from Baseline Heart Rate | 60 minutes
  every one minute after spinal anaesthesia and every five minutes after the delivery of the neonate until the end of the surgery

SECONDARY OUTCOMES:
Sensory blockade | 20 minutes
  Time for onset of sensory block at T4
Motor blockade | 20 minutes
  Time to Bromage 2 and to Bromage 3
Sensory regression | 120 minutes
  Time to two segment regression
Motor block regression | 120 minutes
  Time to Bromage 1 and Bromage 0
Time to maximum effect (Tmax) | 20 minutes
  Time when the motor blockade is complete and sensory blockade is in at the level of T4 dermatome
Time to minimum effect (Tmin) | 120 minutes
  Time to two segment regression of the sensory block (T6) and for motor block regression to Bromage1 and Bromage 0
Nausea | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Scale for nausea (0:no nausea 10:worst possible nausea)
Vomiting | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Number of vomits
Shivering | 0 hours, 2 hours, 4 hours, 8 hours, 24 hours postoperatively
  Yes:shiver No:no shiver
Total ephedrine consumption | 60 minutes
  Total ephedrine consumption intraoperatively
Total phenylephrine consumption | 60 minutes
  Total phenylephrine consumption intraoperatively
Total atropine consumption | 60 minutes
  Total atropine consumption intraoperatively
Neonate Apgar score | 5 minutes
  Apgar score in the 1st and 5th minute after delivery of the neonate
Umbilical cord ph | 15 minutes
  Umbilical cord ph after delivery
Need for administration of antiemetic agent | 90 minutes
  Need for administration of antiemetic agent intraoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieio Hospital, University of Athens, Athens, Attica, Greece